CLINICAL TRIAL: NCT03270852
Title: Enhanced Reality for Hemiparetic Arm in the Stroke Patients; Randomized Case-controlled Clinical Trial for Efficacy
Brief Title: Enhanced Reality for Hemiparetic Arm in the Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ulsan University Hospital (Other)
Responsible Party: Principal Investigator, Chang Ho Hwang, Principal Investigator, Ulsan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: chhwang8
Record Dates: First submitted 2017-08-30; First posted 2017-09-01 (Actual); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Stroke; Paresis; Mirror Movement
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced reality (Experimental): Patients are provided with occupational therapy and physical therapy (task-oriented OT 30 min, FES 20 min) daily for 50 minutes.
  ER therapy is provided 2 times a day for 10 minutes for 2 weeks (10 days of treatment week), except for time of installation, calibration, and 3 minute breaks.
  Interventions: Device: Enhanced reality
- No Enhanced reality (Active Comparator): Patients are provided with occupational therapy and physical therapy (task-oriented OT 30 min, FES 20 min) daily for 50 minutes.
  Interventions: Other: No Enhanced reality

INTERVENTIONS:
Device: Enhanced reality — This prototype is developed by investigators for the first time so that it have no trademark or manufacturer name yet.
  The patient sits facing the horizontal desk with the ER therapy device, and then raises the wrist joint to the fixed base. The hand, wrist, and distal forearm to be treated are positioned below the ER medical camera so that the wrist is visible on the screen. Fix the wrist and wrist joint using Velcro. When treating the distal forearm, detach the wrist fixing Velcro.
  Arms: Enhanced reality
Other: No Enhanced reality — Identical rehabilitation without enhanced reality
  Arms: No Enhanced reality

SUMMARY:
The researchers found that enhanced reality developed for the first time in the word by us had a synergistic or additive effect on brain plasticity in patients without central nervous system injury. The aim of this study is to determine the validity and feasibility of enhanced reality in hemiparetic arm in the stroke patients with central nervous system injury.

DETAILED DESCRIPTION:
Pre-interventional evaluation; within 1 day of initiation of the intervention; 10 days after initiation of the intervention; 30 days after termination of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Arm motor Fugl-Mayer scale; wrist/hand subscales ≥ 2-20
* 9-hole pegboard ; ≥ 25% of contra-lateral hand

Exclusion Criteria:

* Alexander apraxia scale ≤2
* NIH stroke scale question Ia-c ≥1
* Nottingham sensory scale; <75% of contra-lateral hand
* Ashworth scale ≥3
* NIH stroke scale question IX ≥2
* Beck depression inventory ≥21
* Significant upper extremity disease causing hand or below elbow dysfunction
* Visual disturbance
* Refusal of participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2019-06-13 (Actual); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Change of Jebsen Taylor test | 1 day before the initiation of intervention, 10 day after the initiation of intervention, and 30 days after termination of treatment
  Jebsen-Taylor Hand Function Test

SECONDARY OUTCOMES:
Change of Arm motor Fugl-Mayer scale | 1 day before the initiation of intervention, 10 day after the initiation of intervention, and 30 days after termination of treatment
  Arm motor Fugl-Mayer scale; wrist & hand/proximal arm

OTHER OUTCOMES:
Change of Ashworth scale | 1 day before the initiation of intervention, 10 day after the initiation of intervention, and 30 days after termination of treatment
  Ashworth scale; wrist/ elbow
Change of 9-hole pegboard | 1 day before the initiation of intervention, 10 day after the initiation of intervention, and 30 days after termination of treatment
  9-hole pegboard
Change of Stroke impact scale | 1 day before the initiation of intervention, 10 day after the initiation of intervention, and 30 days after termination of treatment
  Stroke impact scale, hand function
Change of Grasp force in Newtons | 1 day before the initiation of intervention, 10 day after the initiation of intervention, and 30 days after termination of treatment
  Grasp force in Newtons
Change of Active range of motion of wrist joint | 1 day before the initiation of intervention, 10 day after the initiation of intervention, and 30 days after termination of treatment
  range of motion of the wrist joint
Change of Korean-modified Barthel index | 1 day before the initiation of intervention, 10 day after the initiation of intervention, and 30 days after termination of treatment
  Korean version-Modified Barthel Index
Change of motor evoked potential of abdutor pollicis brevis | 1 day before the initiation of intervention, 10 day after the initiation of intervention, and 30 days after termination of treatment
  Motor Evoked Potential

CONTACTS AND LOCATIONS:
Overall Officials: Chang Ho Hwang, M.D., Ph.D., Study Director — Ulsan University Hospital
Locations (1):
- Ulsan University Hospital, Ulsan, South Korea

IPD SHARING:
Plan to Share IPD: No